CLINICAL TRIAL: NCT01511172
Title: Effect on Glycemic Control of Individual Maximum Effective Dose of NNC 90-1170 as Add on Therapy to Metformin Compared to Monotherapy of NNC 90-1170 or Metformin or a Metformin-SU Combination Therapy in Patients With Type 2 Diabetes. A Double-blind, Double-dummy, Randomised, Parallel-group, Dose Titration Study With an Open Labelled OHA Arm
Brief Title: Effect of Liraglutide as add-on to Metformin Compared to Either Liraglutide or Metformin Alone, or to a Combination of Metformin and a SU (Sulphonylurea) Agent in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1499
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NNC 90-1170 + Met (Experimental)
  Interventions: Drug: liraglutide; Drug: metformin
- NNC 90-1170 + Met placebo (Experimental)
  Interventions: Drug: placebo
- Met + NNC 90-1170 placebo (Placebo Comparator)
  Interventions: Drug: metformin; Drug: placebo
- Met + Glim (Active Comparator)
  Interventions: Drug: metformin; Drug: glimepiride

INTERVENTIONS:
Drug: liraglutide — Individually adjusted dose, maximum 2.0 mg. Injected subcutaneously
  Arms: NNC 90-1170 + Met
Drug: metformin — 1000 mg daily, administered orally
  Arms: Met + Glim; Met + NNC 90-1170 placebo; NNC 90-1170 + Met
Drug: placebo — Metformin placebo administered orally. 1000 mg daily
  Arms: NNC 90-1170 + Met placebo
Drug: placebo — NNC 90-1170 placebo. Individually adjusted dose, maximum 2.0 mg. Injected subcutaneously
  Arms: Met + NNC 90-1170 placebo
Drug: glimepiride — Individually adjusted dose, administered orally
  Arms: Met + Glim

SUMMARY:
This trial is conducted in Europe and Oceania. The aim of this trial is to assess the effect on glycemic control of NNC 90-1170 (liraglutide) added to metformin compared to metformin given alone in subjects with type 2 diabetes previously treated with OHAs (oral hypoglycaemic agents).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes and treated with at least 50 % of maximum dose(s) of OHA(s) for at least three months
* Duration of type 2 diabetes diagnosis at least one year
* HbA1c 8.0-13.0%, both inclusive
* Body Mass Index (BMI) between 25-40 kg/m^2, both inclusive.

Exclusion Criteria:

* Current treatment with thiazolidinediones or insulin initiated within the last four months prior to trial
* Impaired liver function
* Impaired renal function
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Cancer or any clinically significant disease or disorder, except for conditions associated to the type 2 diabetes, which in the Investigator's opinion could interfere with the results of the trial
* Recurrent major hypoglycaemia as judged by the Investigator
* Known or suspected allergy to trial product or related products
* Use of any drug (except for OHAs), which in the Investigator's opinion could interfere with the glucose level
* Known or suspected abuse of alcohol or narcotics
* Any contraindications to metformin or glimepiride according to the local guidelines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2002-08; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Fasting plasma/serum glucose

SECONDARY OUTCOMES:
Home monitored fasting plasma glucose
Home monitored 7-point glucose profile
Fructosamine
Insulin
C-peptide
HbA1c (glycated haemoglobin A1c)
Weight
Beta-cell function and insulin resistance (HOMA model)
Gastro-intestinal adverse events
Other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (39):
- Australia (4):
  - Novo Nordisk Investigational Site, Daw Park, South Australia
  - Novo Nordisk Investigational Site, Adelaide
  - Novo Nordisk Investigational Site, Ashford
  - Novo Nordisk Investigational Site, Garran
- Novo Nordisk Investigational Site, Vienna, Austria
- Czechia (2):
  - Novo Nordisk Investigational Site, České Budějovice
  - Novo Nordisk Investigational Site, Prague
- Denmark (5):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Frederiksberg
  - Novo Nordisk Investigational Site, Køge
  - Novo Nordisk Investigational Site, Thisted
- France (4):
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Paris
- Germany (7):
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Kaiserslautern
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, Neuss
- Poland (2):
  - Novo Nordisk Investigational Site, Rawa Mazowiecka
  - Novo Nordisk Investigational Site, Zabrze
- United Kingdom (14):
  - Novo Nordisk Investigational Site, Addlestone
  - Novo Nordisk Investigational Site, Aylesbury
  - Novo Nordisk Investigational Site, Barnsley
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Caerleon
  - Novo Nordisk Investigational Site, Camberley
  - Novo Nordisk Investigational Site, Chippenham
  - Novo Nordisk Investigational Site, East Horsley
  - Novo Nordisk Investigational Site, Frome
  - Novo Nordisk Investigational Site, Magherafelt
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Soham
  - Novo Nordisk Investigational Site, Sunbury-on-Thames
  - Novo Nordisk Investigational Site, Yaxley. Peterborough

REFERENCES:
- [Result] Nauck MA, Hompesch M, Filipczak R, Le TD, Zdravkovic M, Gumprecht J; NN2211-1499 Study Group. Five weeks of treatment with the GLP-1 analogue liraglutide improves glycaemic control and lowers body weight in subjects with type 2 diabetes. Exp Clin Endocrinol Diabetes. 2006 Sep;114(8):417-23. doi: 10.1055/s-2006-924230. PMID 17039422
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com